CLINICAL TRIAL: NCT00710814
Title: Effects of Leptin on Body Weight and Neuroendocrine Axes After Gastric Bypass
Brief Title: Trial of Leptin Administration After Roux-en-Y Gastric Bypass
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); Amylin Pharmaceuticals, LLC. (Industry); National Center for Research Resources (NCRR) (NIH)
Responsible Party: Principal Investigator, Judith Korner, Associate Professor of Medicine, Columbia University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: AAAC6692; R21DK081050 (NIH); UL1RR024156 (NIH)
Record Dates: First submitted 2008-07-01; First posted 2008-07-04 (Estimated); Results first posted 2015-11-16 (Estimated); Last update posted 2015-11-16 (Estimated); Status verified 2015-10

CONDITIONS: Overweight
Keywords: Roux-en-Y gastric bypass; Leptin; Bariatric surgery; Overweight after Roux-en-Y gastric bypass surgery
MeSH Terms: conditions — Overweight | interventions — Leptin; metreleptin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Leptin - Placebo (Experimental): Leptin self-administered subcutaneously twice each day for 16 weeks, then Placebo for 16 weeks.
  Interventions: Drug: Leptin; Other: Placebo
- Placebo - Leptin (Placebo Comparator): Placebo self-administered subcutaneously twice each day for 16 weeks, then Leptin for 16 weeks.
  Interventions: Drug: Leptin; Other: Placebo

INTERVENTIONS:
Drug: Leptin — Leptin self-administered subcutaneously at 0.05 mg/kg body weight twice each day
  Other Names: metreleptin
Other: Placebo — Sterile water equal in volume to that of the metreleptin dose calculated for each individual self-administered subcutaneously twice each day

SUMMARY:
This is a pilot and feasibility study to examine a novel intervention using leptin in weight-reduced individuals who have undergone bariatric surgery but still remain obese. Leptin, a peptide hormone secreted from adipose tissue, is a regulator of food intake and energy expenditure. Administration of leptin resulted in profound weight reduction in the few reported cases of obese individuals with genetic leptin deficiency. However, most obese people have increased leptin levels. Such individuals are said to be in a "leptin-resistant" state, whereby administration of physiological concentrations of leptin are ineffective at producing significant weight reduction. Roux-en-Y gastric bypass surgery (RYGBP) is more effective than diet alone in producing long-term reduction of body weight. Yet even after surgery there is a plateau in weight loss though the individual may still be obese and have or be at risk for obesity related morbidities. The investigators have shown that plasma leptin levels are significantly lower in women after RYGBP compared with BMI-matched controls. This state of relative hypoleptinemia or leptin insufficiency suggests that post-RYGBP individuals may be in a "leptin-sensitive" state and, thus, would undergo further weight loss when administered doses of leptin that would not normally result in significant weight reduction. This study will examine the effects of leptin administered by self-injection twice per day on body weight and endocrine function. All individuals will received leptin and placebo and different times during the 34 week study period.

DETAILED DESCRIPTION:
Metreleptin will be self-administered by subcutaneous injection at 0.05 mg/kg body weight twice per day (i.e. at 8 am and 8 pm). This dose was chosen because it would not be expected to cause substantial weight loss in an obese non-surgical population, nor should it incur any substantial injection site reactions. Subjects will receive a demonstration of dose preparation and injection in addition to written instructions with visual aides. After the run-in period, subjects will demonstrate their preparation and injection technique. Placebo injections will consist of sterile water equal in volume to that of the metreleptin dose calculated for each individual. Subjects will be instructed to continue with their current level of physical activity. At week 16, each subject will cross-over to the alternate treatment for an additional 16 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Women ages 25-65 years who are 18 months to 15 years Roux-en-Y gastric bypass
* Current BMI of 28-50 kg/m2 and a percent total body weight loss from highest pre-surgical weight of >20% and <45%
* Must live in the vicinity of New York City to comply with 11 study visits over 34 weeks
* Must be willing to self-inject study drug twice per day

Exclusion Criteria:

* Diabetes
* History of plastic surgery

Ages: 25 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2008-04; Primary Completion 2012-08 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Judith Korner, MD,PhD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Medical Center, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Leptin-Placebo: Leptin self-administered subcutaneously twice each day for 16 weeks, then Placebo for 16 weeks.
- Placebo-Leptin: Placebo self-administered subcutaneously twice each day for 16 weeks, then Leptin for 16 weeks.
Period: Overall Study
Arm/Group | Leptin-Placebo | Placebo-Leptin
Started | 15 | 16
Completed | 14 | 13
Not Completed | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Leptin - Placebo | Placebo - Leptin | Total
Number analyzed (Participants) | 15 | 16 | 31
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 15 | 16 | 31
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: Years] | 50.93 [42 to 61] | 42.76 [29 to 56] | 47 [29 to 61]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 16 | 31
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 15 | 16 | 31

OUTCOME MEASURES:

1. Primary Outcome: Weight Change (in kg.) After Each Intervention
Description: For the Leptin Intervention, 16 week values were compared to baseline for those who received Leptin in the first period, and 32 week values were compared to 16 week values in those who received Leptin in the second period.
  For the Placebo Intervention, 16 week values were compared to baseline for those who received Placebo in the first period, and 32 week values were compared to 16 week values in those who received Placebo in the second period.
Time Frame: 0 weeks, 16 weeks and 32 weeks
Measure: Mean (95% Confidence Interval); unit: kg weight change
Groups:
- Leptin Intervention: Participants in the Leptin-Placebo arm were randomized to first receive Leptin for the first 16 weeks, and participants in the Placebo-Leptin arm were randomized to receive Leptin for the second 16 weeks.
  Both Leptin and placebo were self-administered subcutaneously twice per day.
- Placebo Intervention: Participants in the Placebo-Leptin arm were randomized to receive placebo for the first 16 weeks, and participants in the Leptin-Placebo arm were randomized to receive placebo for the second 16 weeks.
  Both Leptin and placebo were self-administered subcutaneously twice per day.
Arm/Group | Leptin Intervention | Placebo Intervention
Number analyzed (Participants) | 27 | 27
kg weight change | -0.39 [-1.08 to 0.30] | 0.02 [-1.47 to 1.51]

ADVERSE EVENTS:
Time Frame: 32 Weeks
Groups:
- Leptin Intervention: This group "Leptin Intervention" inlcudes the adverse events that were observed while the subjects in either crossover arms when they received Leptin only.
- Placebo Intervention: This group "Placebo Intervention" inlcudes the adverse events that were observed while the subjects in either crossover arms when they received Placebo only.
Arm/Group | Leptin Intervention | Placebo Intervention
Serious Adverse Events (participants affected / at risk) | 0/27 | 0/27
Other Adverse Events (participants affected / at risk) | 9/27 | 4/27
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Leptin Intervention (N=27) | Placebo Intervention (N=27)
Itchiness and bruising at injection site (Skin and subcutaneous tissue disorders) | 9 (9) | 0 (0)
Bruising at injection site (Skin and subcutaneous tissue disorders) | 0 (0) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes